CLINICAL TRIAL: NCT03289195
Title: A Prospective Study To Evaluate The Accuracy Of Percutaneous Breast MRI Biopsy In Diagnosing A Pathologic Complete Response Following Neoadjuvant Chemotherapy
Brief Title: Evaluate The Accuracy Of Breast MRI Biopsy In Diagnosing A Complete Tumor Response For Some Women Following Neoadjuvant Chemotherapy For Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-390
Record Dates: First submitted 2017-09-19; First posted 2017-09-20 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: MRI; Biopsy; 17-390
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This prospective single institution pilot study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI biopsy (Experimental): All patients enrolled will have had complete MR imaging response post Neoadjuvant Chemotherapy (NAC) and will undergo percutaneous MR guided biopsy.
  Interventions: Procedure: MRI Biopsy

INTERVENTIONS:
Procedure: MRI Biopsy — Patient will undergo percutaneous MR guided biopsy by study Breast Radiologist within 0-60 days of completing NAC.

SUMMARY:
The purpose of this study is to test the ability of a breast MRI biopsy to accurately diagnose a complete tumor response to the neoadjuvant chemotherapy (NAC) that the patient just finished. Numerous studies have shown that MRI has the highest accuracy for diagnosing a complete tumor response. The investigator wants to see if in a certain group of women who's breast cancer is no longer visible on the post-treatment MRI that the biopsy specimens from a MRI guided biopsy will accurately diagnose a complete tumor response to treatment which may in the future make breast surgery unnecessary in some women.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 years or older
* Confirmed histologic diagnosis of operable HER2 overexpressing (ER<10%, PR<10%, and HER2 2+ or FISH amplified) OR triple negative (ER<10%, PR<10%, and HER2 0/1+ or 2+/FISH not amplified) OR ER positive invasive ductal or invasive lobular breast cancer including MSKCC pathology confirmation
* Operable breast cancer treated with NAC undergoing either breast conservation or total Mastectomy who have had a post-NAC clinical bilateral breast MRI demonstrating a complete imaging response, which is defined as no residual tumor enhancement.
* No indication of distant metastases (M0)
* Tumor site amenable to MRI guided biopsy as determined by the radiologist
* Definitive surgery being performed at MSKCC within within 0-60 days of completing NAC
* ECOG performance status score of 0 to ≤ 2 and or KPS performance status score of 80% to 100%
* Women of childbearing potential (WOCBP) must not be pregnant.
* Women must not be breastfeeding
* Willing and able to provide informed consent and adhere to the study visit schedule and plan as specified in this protocol

Exclusion Criteria:

* Medical history and concurrent disease:

  * Prior history of treated breast cancer
  * Any underlying medical or psychiatric conditions, which in the opinion of the investigator, will make performing the study intervention hazardous or obscure the interpretation of the results
* Prohibited Treatments and/or Therapies:

  * Prior history of breast cancer surgery and/or radiotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Breast Cancer
Enrollment: 31 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
estimate the negative predictive value (NPV) of a percutaneous MRI biopsy | 2 years
  In this context NPV is defined as the number of true negatives (biopsy negative, i.e., no disease found on the percutaneous biopsy and pCR) divided by the number of all biopsy negatives. While NPV is of primary interest we will also estimate positive predictive value, sensitivity, and specificity of the biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Sutton, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (All Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Suffolk-Commack (All Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Rockville Centre, New York

REFERENCES:
- [Derived] Sutton EJ, Braunstein LZ, El-Tamer MB, Brogi E, Hughes M, Bryce Y, Gluskin JS, Powell S, Woosley A, Tadros A, Sevilimedu V, Martinez DF, Toni L, Smelianskaia O, Nyman CG, Razavi P, Norton L, Fung MM, Sedorovich JD, Sacchini V, Morris EA. Accuracy of Magnetic Resonance Imaging-Guided Biopsy to Verify Breast Cancer Pathologic Complete Response After Neoadjuvant Chemotherapy: A Nonrandomized Controlled Trial. JAMA Netw Open. 2021 Jan 4;4(1):e2034045. doi: 10.1001/jamanetworkopen.2020.34045. PMID 33449096
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm